CLINICAL TRIAL: NCT05396482
Title: Assesment of Hearing in Patients With Vestibular Migraine
Brief Title: Assesment of Hearing in Patients With Vestibular Migra
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rahma Alaa Kamel (Other)
Responsible Party: Sponsor-Investigator, Rahma Alaa Kamel, Rahma Alaa, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Rahma93
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Vestibular Migraine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with vestibular migraine and their relative
  Interventions: Diagnostic Test: Pure tone audiometer

INTERVENTIONS:
Diagnostic Test: Pure tone audiometer — Pure tone audiometer
  Other Names: Otoacustic emission

SUMMARY:
Evaluation of hearing in patients with vestibular migraine

ELIGIBILITY:
Inclusion Criteria:

* vertigo

Exclusion Criteria:

* hypertension

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with vestibular migraine
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-18 (Estimated)

PRIMARY OUTCOMES:
Pathology | 2 years
  For vestibular migraine

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt